CLINICAL TRIAL: NCT04897867
Title: CoolSculpting® Elite: Multi-Country Study to Evaluate Patient Satisfaction for Non-Invasive Fat Reduction in Abdomen, Flanks, Upper Arms, Inner Thighs, Outer Thighs and Submental Area
Brief Title: CoolSculpting® Elite for Non-Invasive Fat Reduction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-MA-PLS-0647
Record Dates: First submitted 2021-05-14; First posted 2021-05-24 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Non-invasive Fat Reduction
Keywords: Fat Reduction Non-invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CoolSculpting® Elite System (Experimental): Participants received up to two CoolSculpting® Elite treatment sessions for the abdomen and flanks plus optional additional body areas 8 weeks apart. At the investigator's discretion, per treatment session, up to 8 treatment cycles were performed for the midsection, and if applicable, up to 2 treatment cycles for the submental area, up to 4 cycles to upper arms, and up to 4 cycles each to inner and/or outer thighs.
  Interventions: Device: CoolSculpting® Elite System with CoolSculpting® Elite applicators

INTERVENTIONS:
Device: CoolSculpting® Elite System with CoolSculpting® Elite applicators — A treatment session is comprised of timed segments of cooling (treatment cycles) followed by 2 minutes of manual massage.

SUMMARY:
This study aims to generate data that conveys participant's experiences such as their satisfaction with treatment delivered by the redesigned CoolSculpting® Elite system for non-invasive fat reduction in the midsection area (abdomen and flanks) in addition to optional body areas of upper arms, inner thighs, outer thighs and/or submental area. By doing this, the study will provide insights for doctors to better inform participants about the expected outcomes when one or more body areas are considered for treatment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Participant must be in good health as determined by medical history, physical examination, vital signs, and investigator's judgment, including no known active pandemic infection.
* Participant has clearly visible and palpable fat in the abdomen and flanks, and participant may also be assessed for visible and palpable fat in one or more of the following body areas: left and right lower aspects of the upper arms, left and right inner thigh, left and right outer thigh, or submental area, which in the investigator's opinion is appropriate for and may benefit from treatment.
* Participant has a BMI of ≥ 18.5 and < 30. BMI is defined as weight in kilograms divided by height in meters squared (kg/m2).
* Participant agrees to maintain weight (ie, within 5% of body weight) by not making any changes in diet or exercise routine during the course of the study.
* Participant agrees to have photographs taken of the treatment area(s) during the scheduled time periods.

Exclusion Criteria:

* Participant has a history of an invasive fat reduction procedure (eg, liposuction, surgery, lipolytic agents, etc) within or adjacent to the area being considered for treatment.
* Participant has implants (eg, breast implants) in or immediately adjacent to the area of intended treatment.
* Participant has a history of prior surgery or scar tissue related to the area being considered for treatment.
* Participant has a known history of cryoglobulinemia, cold urticaria, cold agglutinin disease, or paroxysmal cold hemoglobinuria.
* Participant has a known sensitivity to cold or has any condition with a known response to cold exposure that limits blood flow to the skin, such as cold urticaria, Raynaud's disease, or chilblains (pernio).
* Participant with a clinically significant bleeding disorder, or concomitant use of blood thinners, or is taking any medication that, in the investigator's opinion, may significantly increase the participant's risk of bruising or bleeding.
* Participant has a history of carpal tunnel syndrome, compartment syndrome, or deep vein thrombosis in the upper or lower extremities (only applicable for participants receiving treatment to the upper arms or thighs).
* Participant is currently taking or has taken diet pills or weight control supplements within the past 6 months.
* Participant has any skin conditions, such as moderate to excessive skin laxity, open wound, or scars, and active infection, eczema, dermatitis or rashes in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks are not an exclusion).
* Participant has an active implanted device such as a pacemaker, defibrillator, drug delivery system, or any other metal-containing implant, within or adjacent to the area being considered for treatment.
* Participant (WOCBP- woman of childbearing potential) is pregnant or intending to become pregnant in the next 3 to 6 months and does not agree to use reliable contraception during the study.
* Participant is lactating or has been lactating in the past 6 months.
* Participant is unable or unwilling to comply with the study requirements.
* Participant is currently enrolled in a clinical study of any unapproved investigational device, investigational product, or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Participant has any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the participant's response or the integrity of the data or would pose an unacceptable risk to the participant.
* Participant has had a non-invasive fat reduction and/or body contouring procedure in the area(s) of intended treatment within the past 12 months.
* Participant needs to administer, or has a known history of subcutaneous injections, into the area(s) of intended treatment (eg, cortisone, heparin, insulin) within the past 6 months.
* Participant with known sensitivity or allergy to fructose, glycerin, isopropyl alcohol, or propylene glycol.
* Participant has impaired peripheral circulation in the area to be treated.
* Participant has neuropathic disorders such as post-herpetic neuralgia or diabetic neuropathy.
* Participant has impaired skin sensation in or immediately adjacent to the treatment area(s).
* Participant has a history of hernia in or immediately adjacent to the treatment area(s).
* Participant diagnosed with a systemic fibrosing disease or fibrosis in the area intended or adjacent to the area to be treated.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (8):
- United States (4):
  - Laser & Skin Surgery Medical group, Inc /ID# 239112, Sacramento, California
  - Cosmetic Laser Dermatology /ID# 239110, San Diego, California
  - Cosmetic Laser Dermatology /ID# 239111, San Diego, California
  - Laser & Skin Surgery Center of New York /ID# 239113, New York, New York
- Centre Laser International de la Peau /ID# 239117, Paris, France
- Bodenseeklinik /Id# 239155, Lindau, Germany
- Halley Medical Aesthetics /ID# 239124, Singapore, Singapore
- Akademikliniken /ID# 239120, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CoolSculpting® Elite System
Started | 110
Safety Population (Safety Population consisted of all enrolled participants who received at least one cryolipolysis treatment cycle (started or completed).) | 110
Received Treatment in Session 2 | 100
Evaluable Population 1 (Evaluable Population 1 consisted of all participants who completed the cryolipolysis treatment plan to the midsection and completed the Cryolipolysis Satisfaction Questionnaire (CSQ)-Midsection Item #1 at 12 weeks after the final treatment session and who do not have any significant protocol deviation or violation.) | 96
Evaluable Population 3 (Evaluable Population 3 consisted of all participants who completed the cryolipolysis treatment plan for any body areas (Midsection, Upper Arms, Inner Thighs, Outer Thighs and Submental Area) and do not have any significant protocol deviation or violation.) | 107
Completed | 99
Not Completed | 11
Not completed — Withdrawal of Consent | 1
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 7
Not completed — Reason not Specified | 2

BASELINE CHARACTERISTICS:
Population: Safety Population consisted of all enrolled participants who received at least one cryolipolysis treatment cycle (started or completed).
Arm/Group | CoolSculpting® Elite System
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed is the number of participants at sites in US and Singapore as race and ethnicity were collected only at these sites.
  Participants
    number analyzed (Participants) | 79
    Hispanic or Latino | 7
    Not Hispanic or Latino | 71
    Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Number analyzed is the number of participants at sites in US and Singapore as race and ethnicity were collected only at these sites.
  Participants
    Race: number analyzed (Participants) | 79
    Race: Black or African American | 3
    Race: Chinese | 11
    Race: Middle Eastern | 1
    Race: Taiwanese | 1
    Race: White or Caucasian | 61
    Race: Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With "Satisfied" or "Very Satisfied" on Item #1 for the CSQ (Cryolipolysis Satisfaction Questionnaire) - Midsection
Description: The CSQ-Midsection is a 2-item Patient-reported Outcome (PRO) instrument that measures participant's satisfaction with CoolSculpting® treatment of the midsection (abdomen and flanks). Participants were asked to rate their satisfaction with the results of the fat-reduction procedure on a 5-item scale ranging from Very satisfied to Very dissatisfied.
Time Frame: 12 weeks after the final treatment session (measured at Week 12 for participants who received 1 treatment session or Week 20 for participants who received 2 treatment sessions)
Population: Evaluable Population 1 consisted of all participants who completed the cryolipolysis treatment plan to the midsection and completed the Cryolipolysis Satisfaction Questionnaire (CSQ)-Midsection Item #1 at 12 weeks after the final treatment session and who do not have any significant protocol deviation or violation.
Measure: Number; unit: percentage of participants
Arm/Group | CoolSculpting® Elite System
Number analyzed (Participants) | 96
percentage of participants | 83.3

2. Primary Outcome: Numbers of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Adverse Device Effects (TEADEs); Treatment Emergent Serious Adverse Events (TESAEs), Serious Adverse Device Effects (SADEs), and Unanticipated TEAEs or ADEs
Description: An AE will be considered a TEAE if the AE began or worsened (increased in severity or became serious) on or after the date (and time, if known) of the first dose of study intervention. An AE will be considered a TESAE if it is a TEAE that additionally meets any SAE criterion. TEADE is defined as any TEAE with a reasonable possibility (Possible, Probable, or Causal relationship) that the event may have been caused by the study device. SADE is an ADE that might have led to any SAE consequences if a suitable action had not been taken or intervention had not been made.
Time Frame: First treatment to Follow-up/Exit Visit (Week 12 + 14 days for those participants who received only 1 treatment session and Week 20 + 14 days for those participants who received 2 treatment sessions)
Population: Safety Population consisted of all enrolled participants who received at least one cryolipolysis treatment cycle (started or completed). AEs are reported separately for each of the two treatment sessions.
Measure: Count of Participants; unit: Participants
Groups:
- CoolSculpting® Elite: Treatment Session 1: Participants who received one CoolSculpting® Elite treatment session for the abdomen and flanks plus optional additional body areas. At the investigator's discretion, up to 8 treatment cycles were performed for the midsection and if applicable, up to 2 treatment cycles for the submental area, up to 4 cycles to upper arms, and up to 4 cycles each to inner and/or outer thighs.
- CoolSculpting® Elite: Treatment Session 2: Participants who received a second CoolSculpting® Elite treatment session for the abdomen and flanks plus optional additional body areas. At the investigator's discretion, up to 8 treatment cycles were performed for the midsection and if applicable, up to 2 treatment cycles for the submental area, up to 4 cycles to upper arms, and up to 4 cycles each to inner and/or outer thighs.
Arm/Group | CoolSculpting® Elite: Treatment Session 1 | CoolSculpting® Elite: Treatment Session 2
Number analyzed (Participants) | 110 | 100
Participants
  Any Treatment-Emergent Adverse Event (TEAE) | 5 | 5
  Any Treatment-Emergent Serious Adverse Event (TESAE) | 0 | 0
  Any Unanticipated Treatment-Emergent Adverse Event (UTEAE) | 0 | 0
  Any Unanticipated Treatment-Emergent Serious Adverse Event (UTESAE) | 0 | 0
  Any Treatment-Emergent Adverse Device Effect (TEADE) | 2 | 4
  Any Treatment-Emergent Serious Adverse Device Effect (TESADE) | 0 | 0
  Any Unanticipated Treatment-Emergent Adverse Device Effect (UTEADE) | 0 | 0
  Any Unanticipated Treatment-Emergent Serious Adverse Device Effect (UTESADE) | 0 | 0

3. Secondary Outcome: Percentage of Participants Who Received Treatment to Abdomen and Flank and One or More Additional Body Areas for Treatment With "Satisfied" or "Very Satisfied" on CSQ-Overall Item 1
Description: The CSQ-Overall is a 1-item Patient-reported Outcome (PRO) instrument that measures the participant's satisfaction with CoolSculpting® Elite treatment when midsection and one or more additional body area were selected for treatment. Participants were asked to rate their satisfaction with the results of the fat-reduction procedure when considering the treated areas using a 5-item scale ranging from Very satisfied to Very dissatisfied.
Time Frame: as for outcome 1
Population: Evaluable Population 3 (N=107) consisted of all participants who completed the cryolipolysis treatment plan for any body areas (Midsection, Upper Arms, Inner Thighs, Outer Thighs and Submental Area) and do not have any significant protocol deviation or violation. Overall number analyzed is the number of participants available for analysis for CSQ-Overall Item 1 (n=53).
Measure: Number; unit: percentage of participants
Arm/Group | CoolSculpting® Elite System
Number analyzed (Participants) | 53
percentage of participants | 83.0

4. Secondary Outcome: Percentage of Participants With "Satisfied" or "Very Satisfied" on Individual Treated Body Areas (Upper Arms, Inner Thighs, Outer Thighs, Fat Under Chin) CSQ Item 1
Description: The CSQ- Upper Arms, CSQ-Inner Thighs, CSQ-Outer Thighs, CSQ-Fat Under Chin are 1-item Patient-reported Outcome (PRO) instruments that measure participant's satisfaction with CoolSculpting® Elite treatment for the optional additional individual body area(s) treated. Participants were asked to rate their satisfaction with the results of the fat-reduction procedure for the optional additional individual body area(s) treated on a 5-item scale ranging from Very satisfied to Very dissatisfied.
Time Frame: as for outcome 1
Population: Evaluable Population consisted of all participants who completed the cryolipolysis treatment plan to one or more additional body areas (Upper Arms, Inner Thighs, Outer Thighs, Submental Area), whether midsection treatment was completed or not, and do not have any significant protocol deviation or violation. Number analyzed for each category is the number of participants with available data for the respective individual body area.
Measure: Number; unit: percentage of participants
Arm/Group | CoolSculpting® Elite System
Number analyzed (Participants) | 58
percentage of participants
  CSQ - Inner Thighs: number analyzed (Participants) | 24
  CSQ - Inner Thighs | 58.3
  CSQ - Outer Thighs: number analyzed (Participants) | 3
  CSQ - Outer Thighs | 33.3
  CSQ - Upper Arms: number analyzed (Participants) | 25
  CSQ - Upper Arms | 88.0
  CSQ - Fat Under Chin: number analyzed (Participants) | 6
  CSQ - Fat Under Chin | 83.3

5. Secondary Outcome: Percentage of Participants With Correct Identification of Baseline vs 12-week Post-final Treatment Images of the Treated Body Area(s) by at Least Two Out of Three Blinded, Independent Reviewers
Description: Success was defined as at least 70% correct identification of the pre-treatment images.
Time Frame: 12 weeks after the final treatment session (measured at Week 12 for participants who received 1 treatment session or Week 20 for participants who recieved 2 treatment sessions)
Population: Evaluable Population 3 (N=107) consisted of all participants who completed the cryolipolysis treatment plan for any body areas (Midsection, Upper Arms, Inner Thighs, Outer Thighs and Submental Area) and do not have any significant protocol deviation or violation. Overall number analyzed is the number of participants evaluable for any of the body areas. Number analyzed for each category are the number of participants evaluable for the respective individual body area.
Measure: Number; unit: percentage of participants
Arm/Group | CoolSculpting® Elite System
Number analyzed (Participants) | 107
percentage of participants
  Midsection: number analyzed (Participants) | 92
  Midsection | 88.0
  Inner Thighs: number analyzed (Participants) | 20
  Inner Thighs | 60.0
  Outer Thighs: number analyzed (Participants) | 3
  Outer Thighs | 100
  Upper Arms: number analyzed (Participants) | 25
  Upper Arms | 80.0
  Submental Area: number analyzed (Participants) | 6
  Submental Area | 66.7

ADVERSE EVENTS:
Time Frame: First treatment to Follow-up/Exit Visit (Week 12 +/- 14 days for those participants who received 1 treatment and Week 20 +/- 14 days for those participants who received 2 treatments)
Description: Safety Population consisted of all enrolled participants who received at least one cryolipolysis treatment cycle (started or completed). The data for adverse events is collected and reported per treatment session received. TEAEs occurred on or after the date of treatment session 1 and before the date of treatment session 2 are counted for treatment session 1; TEAEs occurred on or after the date of treatment session 2 are counted for treatment session 2.
Groups:
- CoolSculpting Elite: Treatment Session 1: Participants who received one CoolSculpting® Elite treatment session for the abdomen and flanks plus optional additional body areas. At the investigator's discretion, up to 8 treatment cycles were performed for the midsection and if applicable, up to 2 treatment cycles for the submental area, up to 4 cycles to upper arms, and up to 4 cycles each to inner and/or outer thighs.
- CoolSculpting Elite: Treatment Session 2: Participants who received a second CoolSculpting® Elite treatment session for the abdomen and flanks plus optional additional body areas. At the investigator's discretion, up to 8 treatment cycles were performed for the midsection and if applicable, up to 2 treatment cycles for the submental area, up to 4 cycles to upper arms, and up to 4 cycles each to inner and/or outer thighs.
Arm/Group | CoolSculpting Elite: Treatment Session 1 | CoolSculpting Elite: Treatment Session 2
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/100
Other Adverse Events (participants affected / at risk) | 5/110 | 5/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoolSculpting Elite: Treatment Session 1 (N=110) | CoolSculpting Elite: Treatment Session 2 (N=100)
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
MEDICAL DEVICE PAIN (General disorders) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT04897867/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04897867/SAP_001.pdf